CLINICAL TRIAL: NCT01540487
Title: Characterisation of Fixed Dose Combination Tablets of Linagliptin 2.5 mg/Metformin 850 mg or Linagliptin 2.5 mg/Metformin 500 mg and Relative Oral Bioavailability Compared With Single Linagliptin 2.5 mg and Metformin 850 mg or 500 mg Tablets Administered Together to Healthy Chinese Male and Female Volunteers in an Open Label, Randomised, Single-dose, Two-way Crossover, Phase I Study
Brief Title: Pharmacokinetics of Fixed Dose Combination (FDC) Tablets of Linagliptin /Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.5
Record Dates: First submitted 2012-02-23; First posted 2012-02-28 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (2):
- linagliptin/metformin(high dose) (Experimental): 24 subjects (12 male and 12 female) will be assigned to 2 treatment sequences. cross-over design was adopted to ensure each patient would take fixed dose combination tablets of linagliptin /metformin (high dose) and single linagliptin and metformin (high dose) tablets single dose in randomized order
  Interventions: Drug: linagliptin/metformin(high dose)
- linagliptin/metformin(low dose) (Experimental): 24 subjects (12 male and 12 female) will be assigned to 2 treatment sequences. cross-over design was adopted to ensure each patient would take fixed dose combination tablets of linagliptin /metformin (low dose) and single linagliptin and metformin (low dose) tablets single dose in randomized order
  Interventions: Drug: Linagliptin/metformin(low dose)

INTERVENTIONS:
Drug: linagliptin/metformin(high dose) — patient would take fixed dose combination tablets of linagliptin /metformin (high dose) and single linagliptin and metformin (High dose) tablets single dose in random order, and each dosage will be separated in 42 days interval.
  Arms: linagliptin/metformin(high dose)
Drug: Linagliptin/metformin(low dose) — patient would take fixed dose combination tablets of linagliptin /metformin (low dose) and single linagliptin and metformin (Low dose) tablets single dose in random order, and each dosage will be separated in 42 days interval.
  Arms: linagliptin/metformin(low dose)

SUMMARY:
The aim of the trial is to assess the relative bioavailability of fixed dose combination tablets of linagliptin and metformin compared to the administration of two single tablets (linagliptin and metformin ) in Chinese subjects. The availability of a fixed dose combination tablet is expected to significantly enhance patients' compliance with antidiabetic treatment., in particular with concern to the frequent polypharmacy in diabetic patients.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.5.86001 Boehringer Ingelheim Investigational Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Lina 2.5mg, Metformin 850mg: All patients receiving Linagliptin 2.5mg and Metformin 850mg.
- Lina 2.5mg, Metformin 500mg: All patients receiving Linagliptin 2.5mg and Metformin 500mg.
Period: Overall Study
Arm/Group | Lina 2.5mg, Metformin 850mg | Lina 2.5mg, Metformin 500mg
Started | 24 | 24
Completed | 23 | 24
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lina 2.5mg, Metformin 850mg | Lina 2.5mg, Metformin 500mg | Total
Number analyzed (Participants) | 24 | 24 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.4) | 28.6 (4.8) | 28.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval 0 to 72 Hours (AUC0-72)
Time Frame: 1 hour (h) prior to drug administration, 20 minutes (min), 40 min, 1 h, 1 h 30 min, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, 24 h, 34 h, 48 h and 72 h thereafter.
Population: Treated Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet: Patients receiving 2.5 mg Linagliptin and 850 mg Metformin as a fixed dose combination (FDC) tablet.
- Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets: Patients receiving 2.5 mg Linagliptin and 850 mg Metformin as single tablets.
- Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet: Patients receiving 2.5 mg Linagliptin and 500 mg Metformin as a fixed dose combination (FDC) tablet.
- Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets: Patients receiving 2.5 mg Linagliptin and 500 mg Metformin as single tablets.
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
nmol*h/L | 248 (14.5) | 251 (15.3) | 266 (22.1) | 264 (23.8)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 99.5, 90% CI 2-sided [94.7 to 104.5]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 100.8, 90% CI 2-sided [95.1 to 106.8]

2. Primary Outcome: Maximum Measured Concentration (Cmax) of Linagliptin.
Time Frame: as for outcome 1
Population: Treated Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
nmol/L | 6.90 (23.1) | 6.81 (18.2) | 7.54 (35.4) | 6.77 (25.9)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 101.9, 90% CI 2-sided [95.4 to 109.0]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 111.4, 90% CI 2-sided [100.4 to 123.5]

3. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval 0 to the Last Quantifiable Concentration (AUC0-tz)
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
ng*h/mL | 11700 (27.9) | 12100 (23.2) | 8240 (20.8) | 8010 (21.3)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 97.0, 90% CI 2-sided [90.6 to 103.8]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusteg gMean ratio = 103.0, 90% CI 2-sided [96.2 to 110.1]

4. Primary Outcome: Maximum Measured Concentration (Cmax) of Metformin
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
ng/mL | 1680 (34.8) | 1780 (26.0) | 1220 (29.1) | 1190 (27.2)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 94.6, 90% CI 2-sided [85.4 to 104.8]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 102.5, 90% CI 2-sided [92.2 to 113.9]

5. Secondary Outcome: Area Under the Concentration Time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity) for Linagliptin
Description: AUC0-infinity is based on predicted last concentration values.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
nmol*h/L | 471 (29.8) | 433 (22.2) | 483 (32.5) | 541 (36.4)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 110.1, 90% CI 2-sided [100.5 to 120.6]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 89.3, 90% CI 2-sided [80.2 to 99.3]

6. Secondary Outcome: AUC(0-infinity) for Metformin
Description: AUC0-infinity is based on predicted last concentration values.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
ng*h/mL | 12200 (25.8) | 12500 (23.0) | 8440 (19.3) | 8210 (20.3)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 98.0, 90% CI 2-sided [92.0 to 104.5]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 102.8, 90% CI 2-sided [97.0 to 109.0]

7. Secondary Outcome: AUC0-tz for Linagliptin
Time Frame: as for outcome 1
Population: Treated Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Number analyzed (Participants) | 23 | 24 | 24 | 24
nmol*h/L | 248 (14.5) | 251 (15.3) | 266 (22.1) | 264 (23.8)
Statistical Analysis 1: Comparison: Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 99.5, 90% CI 2-sided [94.7 to 104.6]
Statistical Analysis 2: Comparison: Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet vs Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets; Test type: Superiority or Other; ANOVA; adjusted gMean ratio = 100.8, 90% CI 2-sided [95.1 to 106.8]

ADVERSE EVENTS:
Time Frame: First treatment with study drug until End-of-Study (which was 7 to 14 days after study drug treatment in Visit 3), i.e. 7 weeks plus 4 to 11 days after first treatment with study drug
Arm/Group | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 2/24 | 0/24 | 2/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linagliptin 2.5 mg, Metformin 850 mg as FDC Tablet (N=23) | Linagliptin 2.5 mg, Metformin 850 mg as Single Tablets (N=24) | Linagliptin 2.5 mg, Metformin 500 mg as FDC Tablet (N=24) | Linagliptin 2.5 mg, Metformin 500 mg as Single Tablets (N=24)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.